CLINICAL TRIAL: NCT01598298
Title: A Randomized Placebo-Controlled Phase III Study of Duloxetine for Treatment of Aromatase Inhibitor-Associated Musculoskeletal Symptoms in Women With Early Stage Breast Cancer
Brief Title: S1202: Duloxetine Hydrochloride for Muscle/Joint Pain in Early-Stage Breast Cancer Receiving Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S1202; S1202 (Other: SWOG); U10CA037429 (NIH); NCI-2012-01960 (Other: NCI)
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Musculoskeletal Complications; Pain
Keywords: estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; pain; musculoskeletal complications
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive duloxetine hydrochloride orally (PO) once daily (QD) on days 1-7, twice daily (BID) on days 8-84, and then QD on days 85-91.
  Interventions: Drug: duloxetine hydrochloride
- Arm II (Placebo Comparator): Patients receive placebo PO QD on days 1-7, BID on days 8-84, and then QD on days 85-91.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: duloxetine hydrochloride — Given PO
  Other Names: NSC-744012
  Arms: Arm I
Other: placebo — Given PO
  Arms: Arm II

SUMMARY:
RATIONALE: Duloxetine hydrochloride may lessen muscle, bone, and joint pain caused by hormone therapy. It is not yet known whether duloxetine hydrochloride is more effective than a placebo in treating patients with muscle, bone, and joint pain caused by hormone therapy.

PURPOSE: This randomized phase III trial studies how well duloxetine hydrochloride works compared to a placebo in treating muscle, bone, and joint pain in patients with early-stage breast cancer receiving hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether daily duloxetine hydrochloride (duloxetine) decreases average joint pain in women with aromatase inhibitor-associated musculoskeletal syndrome (AIMSS), as measured at 12 weeks by the modified Brief Pain Inventory Short Form (BPI-SF).

Secondary

* To assess whether daily duloxetine decreases worst joint pain in women with AIMSS, as measured at 12 weeks by the modified BPI-SF.
* To assess whether daily duloxetine decreases pain interference in women with AIMSS, as measured at 12 weeks by the modified BPI-SF.
* To investigate whether daily duloxetine improves functioning, pain, and stiffness in the knees/hips according to the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) scale. (Exploratory)
* To investigate whether daily duloxetine improves function, pain, and stiffness in the hands according to the Modified Score for the Assessment and Quantification of Chronic Rheumatoid Affections of the Hands (M-SACRAH). (Exploratory)
* To investigate whether daily duloxetine improves functional quality of life as measured by the Functional Assessment of Cancer Therapy-Endocrine Scale (FACT-ES). (Exploratory)
* To investigate whether daily duloxetine improves the proportion of patients reporting changes for the better versus worst as measured by the Global Rating of Change Scale. (Exploratory)
* To investigate whether daily duloxetine decreases analgesic use.
* To investigate whether daily duloxetine increases adherence to, and reduces the discontinuation rate for, aromatase inhibitor (AI) therapy. (Exploratory)
* To assess whether patients receiving duloxetine as compared to placebo have improved depression as measured by the Patient Health Questionnaire (PHQ-9) at Weeks 6 and 12. (Exploratory)
* To explore the relationship between inherited variants in genes responsible for duloxetine metabolism and activity (COMT, HTR3A, SLC6A2, SLC6A4, CYP1A2, CYP2D6) and aromatase (CYP19A1) and change in pain with 12 weeks of treatment. (Exploratory)
* To explore the impact of treatment on serum inflammatory cytokine levels with 12 weeks of treatment at baseline and 12 weeks. (Exploratory)
* To bank blood samples for future correlative analyses. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to baseline pain score (4-6 vs 7-10), and prior taxane use (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive duloxetine hydrochloride orally (PO) once daily (QD) on days 1-7, twice daily (BID) on days 8-84, and then QD on days 85-91.
* Arm II: Patients receive placebo PO QD on days 1-7, BID on days 8-84, and then QD on days 85-91.

Patients complete the modified Brief Pain Inventory Short Form (BPI-SF) questionnaire at baseline and periodically during study treatment. Patients may also complete the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) scale, the Modified Score for the Assessment and Quantification of Chronic Rheumatoid Affections of the Hands (M-SACRAH), the Functional Assessment of Cancer Therapy-Endocrine Scale (FACT-ES), Global Rating of Change Scale, and the patient Health Questionnaire (PHQ-9).

Patients undergo blood sample collection at baseline and periodically during treatment for correlative studies, including biomarker and genetic studies.

After completion of study treatment, patients are followed up for 168 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must be women with histologically confirmed estrogen receptor (ER)- and/or progesterone receptor (PgR)-positive invasive carcinoma of the breast with no evidence of metastatic disease (M0)
* Patients must have completed mastectomy or breast-sparing surgery and must have recovered from all side effects of the surgery
* Patients must have aromatase inhibitor (AI)-associated musculoskeletal symptoms that began or increased after starting AI therapy; new musculoskeletal pain must not be due specifically to fracture or traumatic injury
* Patients must have completed the S1202 Brief Pain Inventory-Short Form (BPI-SF) within 7 days prior to registration; patients must have an "average pain" of at least 4 on the BPI-SF

PATIENT CHARACTERISTICS:

* Patients must be post-menopausal, as defined by at least one of the following:

  * At least 12 months since the last menstrual period
  * Prior bilateral oophorectomy
  * Previous hysterectomy with one or both ovaries left in place (or previous hysterectomy in which documentation of bilateral oophorectomy is unavailable) AND follicle-stimulating hormone (FSH) values consistent with the institutional normal values for the post menopausal state; if patient is under the age of 55, FSH levels must be obtained within 28 days prior to registration OR
  * Have been on LHRH agonist therapy for at least 3 months and estradiol levels drawn within 28 days prior to registration are consistent with the institutional normal values for post-menopausal state.
* Patients must have Zubrod performance status of 0-2
* Patients must have no known allergy or hypersensitivity to duloxetine or any of the inactive ingredients in the matching placebo
* Patients must not have any contraindicated concurrent illnesses listed on the duloxetine package insert including:

  * Current primary psychiatric diagnosis (schizophrenia, psychosis) or suicidal ideation, history of bipolar disorder, or seizure disorder
  * History of alcohol or other substance abuse or dependence within 365 days prior to registration
  * Chronic liver disease
  * End-stage renal disease
  * Uncontrolled narrow-angle glaucoma
  * Clinically significant coagulation disorder
* Creatinine clearance > 30 mL/min
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both within 3 x upper limit of normal
* Total bilirubin within the upper limit of normal
* Patients must be able to complete study questionnaires in English or Spanish
* Patients must not have concurrent medical/arthritic disease that could confound or interfere with evaluation of pain or efficacy including: inflammatory arthritis (rheumatoid arthritis, systemic lupus, spondyloarthropathy, psoriatic arthritis, polymyalgia rheumatica), or cancer involving the bone
* Patients must be willing to submit blood samples for correlative studies; baseline samples must be obtained prior to beginning protocol treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* If patients were treated with chemotherapy and/or radiation therapy, these treatments must be completed at least 28 days prior to study registration
* Concurrent bisphosphonate and trastuzumab therapies are allowed
* Patients should have recovered from all Grade 2 or higher side effects of chemotherapy and/or radiation therapy with the exception of alopecia and peripheral neuropathy
* Patients must currently be taking one of the following aromatase inhibitor (AI) doses for at least 21 days, but no longer than 12 months, prior to registration and plans to continue for at least an additional 180 days after registration

  * Anastrozole (Arimidex®) 1 mg daily
  * Letrozole (Femara®) 2.5 mg daily
  * Exemestane (Aromasin®) 25 mg daily
* Patients must not be taking any contraindicated medications listed on the duloxetine package insert including the following: treatment with phenothiazines, propafenone, flecainide, or linezolid; treatment with monoamine oxidase (MAO)-inhibitor within 14 days prior to registration; or current use of anticoagulation medication (e.g., heparin, warfarin)
* Patients must not require selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephirine reuptake inhibitors (SNRIs), or tricyclic antidepressants during study participation; patients must have been able to taper and discontinue treatment with these medications at least 7 days prior to registration; patients must not have taken duloxetine or milnacipran within 90 days prior to registration
* Patients who are receiving treatment with narcotics, tramadol, gabapentin, and/or pregabalin must have been taking a stable dose for at least 30 days prior to registration

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: N. Lynn Henry, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center; Anne F. Schott, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (714):
- United States (714):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Cancer Center of South Florida-Lake Worth, Lake Worth, Florida
  - The Watson Clinic, Lakeland, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Little Company of Mary Hospital, Evergreen Park, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care-North, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Porter Memorial Hospital, Valparaiso, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Norwood Hospital, Norwood, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren-Bay Region, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Great Lakes Cancer Institute, Clarkston, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Family Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Family Cancer Center-Southhaven, Southaven, Mississippi
  - Baptist Memorial Hospital-Desoto, Southhaven, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Medical Offices West, Norfolk, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Urology Cancer Center PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Alpine Hematology-Oncology, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Reno Oncology Consultants, Reno, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Queens Hospital Center, Jamaica, New York
  - Orange Regional Medical Center, Middletown, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Gaston Hematology and Oncology Associates-Belmont, Belmont, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Gaston Hematology and Oncology Associates, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Cape Fear Cancer Specialists-Leland, Leland, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Carolina Oncology Associates PA, Salisbury, North Carolina
  - Cleveland Hematology and Oncology Associates PC, Shelby, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Marion L Shepard Cancer Center at Vidant Beaufort Hospital, Washington, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Cape Fear Cancer Specialists, Wilmington, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OneHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Holy Redeemer Hospital and Medical Center, Meadowbrook, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center, Williamsport, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Boston Baskin Cancer Center-Bartlett, Bartlett, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Technology University, El Paso, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - IMG Hematology Oncology 8501, Fairfax, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Wheaton Franciscan Healthcare - Saint Joseph, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
https://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- [Derived] Henry NL, Unger JM, Schott AF, Fehrenbacher L, Flynn PJ, Prow DM, Sharer CW, Burton GV, Kuzma CS, Moseley A, Lew DL, Fisch MJ, Moinpour CM, Hershman DL, Wade JL 3rd. Randomized, Multicenter, Placebo-Controlled Clinical Trial of Duloxetine Versus Placebo for Aromatase Inhibitor-Associated Arthralgias in Early-Stage Breast Cancer: SWOG S1202. J Clin Oncol. 2018 Feb 1;36(4):326-332. doi: 10.1200/JCO.2017.74.6651. Epub 2017 Nov 14. PMID 29136387
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Duloxetine: Patients receive duloxetine hydrochloride orally (PO) once daily (QD) on days 1-7, twice daily (BID) on days 8-84, and then QD on days 85-91.
  duloxetine hydrochloride: Given PO
- Arm II: Placebo: Patients receive placebo PO QD on days 1-7, BID on days 8-84, and then QD on days 85-91.
  placebo: Given PO
Period: Overall Study
Arm/Group | Arm I: Duloxetine | Arm II: Placebo
Started | 150 | 149
Patients Evaluable for Primary Endpoint (Patient has an in-window BPI assessment at week 2, 6, or 12.) | 127 | 128
Patients Evaluable for Adverse Events | 138 | 141
Completed | 110 | 108
Not Completed | 40 | 41
Not completed — Not eligible | 5 | 5
Not completed — Adverse Event | 21 | 19
Not completed — Progression/relapse | 0 | 2
Not completed — Withdrawal by Subject | 10 | 15
Not completed — Other reason (not protocol specified) | 4 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Duloxetine | Arm II: Placebo | Total
Number analyzed (Participants) | 145 | 144 | 289
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 83] | 60 [27 to 82] | 60 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 144 | 289
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 140 | 137 | 277
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 17 | 27
  White | 128 | 120 | 248
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Baseline pain score [Count of Participants; unit: Participants] — Baseline pain score is the patient's self-reported average pain at baseline as measured by the BPI-SF question, "Please rate your joint pain by selecting the one number that best describes your joint pain on the AVERAGE". This score ranges from 0 to 10, with higher scores indicating more pain.
  Participants
    4-6 | 110 | 110 | 220
    7-10 | 35 | 34 | 69
Prior taxane use [Count of Participants; unit: Participants]
  No | 68 | 65 | 133
  Yes | 77 | 79 | 156

OUTCOME MEASURES:

1. Primary Outcome: Average Joint Pain According to BPI-SF
Description: Average joint pain according to the Brief Pain Inventory - Short Form (BPI-SF) average pain score (item #4). This item has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine".
Time Frame: Weeks 2, 6, 12, and 24; Week 12 reported
Population: Patients evaluable for primary endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I: Duloxetine | Arm II: Placebo
Number analyzed (Participants) | 127 | 128
units on a scale | 2.9 (2.1) | 3.5 (2.1)
Statistical Analysis 1: Comparison: Arm I: Duloxetine vs Arm II: Placebo; The primary analysis will rely on longitudinal measures of BPI at Weeks 2, 6, and 12 for improved power. Assessment windows of +/- 7 days, +/- 14 days, and +/- 14 days will be allowed for the 2, 6, and 12 week timepoints. The analysis will be performed using mixed models, adjusted for the stratification factors; Test type: Other — Two-sided test at the alpha=0.05 level; p = 0.0002, Mixed Models Analysis — Two-sided p-value; alpha=0.05; Adjusted for the protocol-specified stratification factors (baseline average pain and prior taxane use); Coefficient for treatment term = -0.82, 95% CI 2-sided [-1.24 to -0.40] — The estimation parameter is the model-based coefficient for the treatment term, with placebo as the reference level

2. Secondary Outcome: Worst Joint Pain According to the BPI-SF
Description: Worst joint pain according to the BPI-SF worst pain score (item #2). This item has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine".
Time Frame: Weeks 2, 6, 12, and 24; Week 12 reported
Population: Patients evaluable for primary endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I: Duloxetine | Arm II: Placebo
Number analyzed (Participants) | 127 | 128
units on a scale | 4.0 (2.8) | 4.9 (2.7)
Statistical Analysis 1: Comparison: Arm I: Duloxetine vs Arm II: Placebo; The primary analysis will rely on longitudinal measures of BPI at Weeks 2, 6, and 12 for improved power. Assessment windows of +/- 7 days, +/- 14 days, and +/- 14 days will be allowed for the 2, 6, and 12 week timepoints. The analysis will be performed using mixed models, adjusted for baseline worst pain score and the stratification factors; Test type: Other — Two-sided test at the alpha=0.05 level; p < 0.0001, Mixed Models Analysis — Two-sided p-value; alpha=0.05; Adjusted for baseline worst pain score and the protocol-specified stratification factors (baseline average pain and prior taxane use); Coefficient for treatment term = -1.06, 95% CI 2-sided [-1.57 to -0.55] — The estimation parameter is the model-based coefficient for the treatment term, with placebo as the reference level

3. Secondary Outcome: Pain Interference According to the BPI-SF
Description: Pain interference according to the BPI-SF: this item has a scale of 0 to 10 with 0 indicating "Does not interfere" and 10 indicating "Completely interferes".
Time Frame: Weeks 2, 6, 12, and 24; Week 12 reported
Population: Patients evaluable for primary endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I: Duloxetine | Arm II: Placebo
Number analyzed (Participants) | 127 | 128
units on a scale | 1.9 (2.2) | 2.6 (2.1)
Statistical Analysis 1: Comparison: Arm I: Duloxetine vs Arm II: Placebo; The primary analysis will rely on longitudinal measures of pain interference scores at Weeks 2, 6, and 12 for improved power. Assessment windows of +/- 7 days, +/- 14 days, and +/- 14 days will be allowed for the 2, 6, and 12 week timepoints. The analysis will be performed using mixed models, adjusted for baseline pain interference score and the stratification factors; Test type: Other — Two-sided test at the alpha=0.05 level; p < 0.0001, Mixed Models Analysis — Two-sided p-value; alpha=0.05; Adjusted for baseline pain interference score and the protocol-specified stratification factors (baseline average pain and prior taxane use); Coefficient fro treatment term = -0.95, 95% CI 2-sided [-1.35 to -0.55] — The estimation parameter is the model-based coefficient for the treatment term, with placebo as the reference level

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: Only adverse events and serious adverse events that are possibly, probably or definitely related to study drug are reported.
Arm/Group | Arm II: Placebo | Arm I: Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/138
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/138
Other Adverse Events (participants affected / at risk) | 83/141 | 115/138
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm II: Placebo (N=141) | Arm I: Duloxetine (N=138)
Vertigo (Ear and labyrinth disorders) | 6 | 10
Abdominal pain (Gastrointestinal disorders) | 6 | 11
Constipation (Gastrointestinal disorders) | 9 | 23
Diarrhea (Gastrointestinal disorders) | 10 | 21
Dry mouth (Gastrointestinal disorders) | 20 | 38
Nausea (Gastrointestinal disorders) | 12 | 47
Vomiting (Gastrointestinal disorders) | 2 | 7
Fatigue (General disorders) | 25 | 52
Flu like symptoms (General disorders) | 1 | 12
Pain (General disorders) | 23 | 27
Anorexia (Metabolism and nutrition disorders) | 3 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 31
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 13 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 32
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 8
Dizziness (Nervous system disorders) | 5 | 20
Headache (Nervous system disorders) | 30 | 35
Lethargy (Nervous system disorders) | 1 | 9
Paresthesia (Nervous system disorders) | 10 | 7
Somnolence (Nervous system disorders) | 4 | 14
Tremor (Nervous system disorders) | 0 | 11
Agitation (Psychiatric disorders) | 7 | 10
Insomnia (Psychiatric disorders) | 12 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 13
Hot flashes (Vascular disorders) | 22 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT01598298/Prot_SAP_ICF_000.pdf